CLINICAL TRIAL: NCT04439331
Title: MATCH Treatment Subprotocol U: VS-6063 (Defactinib) in Patients With Tumors With NF2 Loss
Brief Title: Testing VS-6063 (Defactinib) as a Potential Targeted Treatment in Cancers With NF2 Genetic Changes (MATCH-Subprotocol U)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-03368; NCI-2020-03368 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-U (Other: ECOG-ACRIN Cancer Research Group); EAY131-U (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2020-06-18; First posted 2020-06-19 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphoid Cell Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Hematologic Neoplasms; Lymphoma; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (defactinib) (Experimental): Patients receive defactinib PO 400 mg BID on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Defactinib Hydrochloride

INTERVENTIONS:
Drug: Defactinib Hydrochloride — Given PO

SUMMARY:
This phase II MATCH treatment trial identifies the effects of VS-6063 (defactinib) in patients whose cancer has a genetic change called NF2 mutation. Defactinib may block a protein called FAK, which may be needed for cancer cell growth when NF2 mutations are present. Researchers hope to learn if defactinib will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive defactinib hydrochloride (defactinib) orally (PO) 400 mg twice daily (BID) on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

THE MATCH SCREENING TRIAL:

Please see NCT02465060 for information on the MATCH Screening Protocol and applicable documents.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients must have a tumor that harbors an inactivating mutation in NF2
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients with known left ventricular dysfunction must have echocardiogram (ECHO) or a nuclear study (multigated acquisition scan [MUGA] or First Pass) within 4 weeks prior to registration to treatment and must not have left ventricular ejection fraction (LVEF) < institutional lower limit of normal (LLN). If the LLN is not defined at a site, the LVEF must be > 50% for the patient to be eligible
* Patients with history of hypertension should be adequately controlled (blood pressure [BP] < 140/90) with appropriate anti-hypertensive therapy or diet

Exclusion Criteria:

* Patients must not have known hypersensitivity to VS-6063 (defactinib) or compounds of similar chemical or biologic composition
* Patients must not have a history of upper gastrointestinal (GI) bleeding, ulceration, or perforation within 12 months prior to the first dose of study drug
* Patients must not have known history of Gilbert's syndrome
* Patient must not have a known history of stroke or cerebrovascular accident within 6 months prior to the first dose of VS-6063 (defactinib)
* Patients must not have prior treatment with a FAK inhibitor (e.g., VS-6063 [defactinib] or GSK2256098) and must not be participating or have participated in the COMMAND trial of maintenance therapy of VS-6063 (defactinib) versus (vs.) placebo, for mesothelioma
* Patients must not be using drugs or foods that are known potent CYP3A4 or CYP2C9 inhibitors or inducers. Substrates of CYP3A4, 2C9, UGT1A1, P-gp, OATP1B1, and OATP1B3 should be used with caution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David M Jackman, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol U was activated on August 12, 2015. Thirty-five patients were enrolled on EAY131-U between November 19, 2015, and November 8, 2017. Twenty-seven patients were enrolled on the basis of the results from the NCI-MATCH assay and 8 on the basis of the outside assay results.
Pre-assignment Details: Patients whose tumors harbored an inactivating NF2 mutation on next-generation sequencing were assigned to sub-protocol U. The mutation status was determined by an NCI-MATCH approved laboratory for 8 patients in this arm, these cases had to be confirmed to be used in primary analysis.
Period: Overall Study
Arm/Group | Treatment (Defactinib)
Started | 35
Started Protocol Therapy | 33
Eligible, Treated and Mutation Status Confirmed (Primary efficacy analysis set) | 30
Completed | 0
Not Completed | 35
Not completed — Never Start Protocol Therapy | 2
Not completed — Ineligible | 2
Not completed — Mutation Status Not Confirmed | 1
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Disease Progression | 20
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 1
Not completed — Other Complicating Disease | 1

BASELINE CHARACTERISTICS:
Population: Patients who were eligible, started protocol therapy, and had mutation status confirmed at the analysis time were the analyzable patients
Arm/Group | Treatment (Defactinib)
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 61 [20 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 25
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Details about how to define complete response and partial response can be found in the master protocol. 90% two-sided binomial exact confidence interval is calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Defactinib)
Number analyzed (Participants) | 30
percentage of participants | 3.2 [0.17 to 14.9]

2. Secondary Outcome: 6-month Progression Free Survival (PFS)
Description: Progression free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS rate is determined
Population: Eligible, treated and mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Defactinib)
Number analyzed (Participants) | 30
percentage of participants | 22.8 [11.2 to 36.7]

3. Secondary Outcome: Progression Free Survival
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first. Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and mutation status confirmed
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Defactinib)
Number analyzed (Participants) | 30
months | 1.9 [1.8 to 3.6]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All patients enrolled were included in the all-cause mortality analysis. Thirty-three patients were included in the toxicity analysis (excluding two who did not receive treatment).
Arm/Group | Treatment (Defactinib)
All-Cause Mortality (participants affected / at risk) | 29/35
Serious Adverse Events (participants affected / at risk) | 9/33
Other Adverse Events (participants affected / at risk) | 22/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Defactinib) (N=33)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Defactinib) (N=33)
Anemia (Blood and lymphatic system disorders) | 6
Edema limbs (General disorders) | 4
Fatigue (General disorders) | 11
Diarrhea (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 10
Stomach pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 5
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 9
Lymphocyte count decreased (Investigations) | 3
White blood cell decreased (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Hematuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT04439331/Prot_002.pdf
  • Informed Consent Form (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT04439331/ICF_003.pdf